CLINICAL TRIAL: NCT03666611
Title: Supporting Family Carers to People Living With Symptoms of Dementia at Home up to the End of Life: a Retrospective Qualitative Study Using Principles of Grounded Theory
Brief Title: Supporting Family Carers to People Living With Symptoms of Dementia at Home up to the End of Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Sara Yearsley, PhD research assistant, University of Manchester
Other Study IDs: sy
Record Dates: First submitted 2018-09-09; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Family Caregivers
Keywords: Dementia; End of Life; Palliative
MeSH Terms: conditions — Dementia; Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a qualitative study that will seek to gain further understanding of the support needs of family carers to people living with symptoms of dementia up to the end of life.

Family carers are friends, family members or neighbours who provide informal unpaid care to someone with symptoms of dementia. The experience of providing this care may result in family carers developing unmet needs that impact adversely on their total wellbeing. This research is potentially beneficial because little is known about the specific physical, psychological, spiritual and social needs family carers to people dying with dementia may develop.

It is a priority of the UK government and the NHS to better support family carers. The government published guidelines calling on healthcare professionals to assess and address carer needs, but the evidence base for family carers to people with symptoms of dementia is limited. Findings from this study could guide healthcare professionals when they conduct clinical assessments of carer needs.

Each participant to this study will be invited to attend a semi-structured interview at a venue of their choice where they will talk about their experiences of providing care. Participants must have provided informal, unpaid care to a friend, neighbour or family member with symptoms of dementia at home, including within the last twelve months of that person's life. This is a retrospective study so only former family carers will be eligible to participate. Participants must also be over the age of eighteen, be able to communicate in English and have capacity to give informed consent.

This research study is being funded by the National Institute for Health Research (NIHR) Collaboration for Leadership in Applied Health Research and Care (CLAHRC) as part of their Research Capacity in Dementia Care Pilot Programme, which is exploring issues relating to dementia care provision.

DETAILED DESCRIPTION:
This study will seek to explore the experiences of former family carers who supported someone living with symptoms of dementia at home up to their death.

The principal research objective will be to identify the support needs common to this group of family carers. The study will explore the main factors that bring about these needs and it will aim to determine whether a carer's needs change as the health of the person receiving care deteriorates towards the end of life. The study will also seek to learn more about the types of assistance family carers receive from health and social care professionals, family members, friends, neighbours and the voluntary sector.

The principal research objective can be of value because it offers family carers an opportunity to share their personal stories, insights and experiences. Providing this information can increase awareness of the carers' role and indicate why a family carer's total health and wellbeing can decline whilst providing informal support to someone living with symptoms of dementia, especially as the care recipient nears death.

The findings from this study should enable healthcare professionals to conduct more informed assessments of carer capacity and wellbeing. The information collected in this study may also identity interventions that carers felt successfully enhanced their wellbeing and reduced their needs, particularly at the time when the person they cared for approached the end of life.

This study will also consider the effectiveness of the Carer Support Needs Assessment Tool (CSNAT) intervention when used by home-based family carers supporting someone living with symptoms of dementia.

This assessment tool has been designed to identify the needs of family carers to people with a life-limiting health condition. The CSNAT helps these carers to prioritise their needs and seek appropriate solutions. It also enables healthcare professionals to provide more tailored support.

This is a qualitative study. Approximately thirty participants will be recruited and each be asked to take part in a semi-structured interview. The researcher will also record observational data in the form of reflective, contemporary field notes.

People who have provided informal, unpaid care to a friend, neighbour or family member with symptoms of dementia will be asked to participate. The support they have given may have been provided on either a permanent or intermittent basis, however all participants must have had some involvement in the provision of home-based care during the last twelve months of the care recipient's life. This is a retrospective study. The care recipient must have died not less than six months and not more than five years before the interview takes place. All participants must also be over eighteen years of age, be able to communicate in English and have capacity to provide informed consent.

Participants will be recruited with the assistance of health and social care professionals including an Admiral Nurse Manager. Healthcare agencies, charities, community organisations and groups that represent older adults have also been approached. Representatives from these organisations will be asked to send participant recruitment packs to all former family carers listed on their caseloads/databases who meet the inclusion criteria.

Details of the study will be uploaded onto forums of dementia, carer and research-related websites including www.joindementiaresearch.co.uk. The researcher will also request permission to put up informational posters in local community centres including GP practices. The posters will include the researcher's contact details so anyone who wishes to receive more information about the study can do so. The researcher will attend meetings of local support groups to raise awareness about the study, answer questions and distribute participant recruitment packs to possible volunteers. In addition, potential participants who express an interest in the research study via word of mouth will also be sent participant recruitment packs.

The participant recruitment packs will include an introductory letter and participant information sheet. Anyone who is interested in participating or who would like to discuss the study in more detail with the researcher can complete an expression of interest form and return it in a stamped addressed envelope. The form and envelope will be included in the participant recruitment packs.

The researcher will telephone those who return a reply form in order to discuss their voluntary participation in the study, provide them with details of what they will be asked to do, ensure they meet the inclusion criteria and answer any questions before scheduling an interview date and location. All interviews will be conducted at least forty-eight hours following this telephone conversation to give participants opportunity to reflect on their decision to take part. No further contact will be attempted with those who do not respond after receiving a participant recruitment pack.

Each participant will be interviewed on one occasion by the researcher in a location of their choice. They will be informed that the researcher will be happy to interview them in their own homes if this is convenient. Participants will not be paid, however any reasonable transport, refreshment or sundry costs will be met by the researcher. Before signing the consent form, each participant will be informed that they can decline to answer any question or withdraw from the research study at any time. They will be assured that their healthcare treatment will not be affected in any way if they do withdraw from the study.

During the interview, participants will be asked to share their experiences of caring for a person with symptoms of dementia. A broad interview protocol will be used to guide the semi-structured interview. The interview will focus on topics including the participants' needs, the factors that generated the needs and also how the needs changed as the person the participant cared for neared the end of life. Participants will be prompted to reflect on the support they received from others. There will, however, be some flexibility to the interview's underlying structure. The interview should feel conversational in tone and participants will be encouraged to talk openly and raise issues that they consider important and relevant.

During the interview, participants will also be shown a copy of the Carer Support Needs Assessment Tool (CSNAT). A large print copy of the tool will be provided for any participant with poor eyesight. Participants will be asked for their thoughts on the tool and its ease of use.

The researcher will telephone all participants who gives prior. signed consent in the week following their interviews to ask them to share any further thoughts on the issues discussed. It has been found that participants often reflect on their responses to interview questions after the event and many recall insightful additional information once the interview has concluded. Capturing this thoughtful, valuable data can add to the quality and depth of the study. Participants will be informed prior to giving consent that the telephone call will be recorded and anonymised quotes may be used by the researcher in academic articles or in her final thesis. Participants will be reminded of this at the start of the telephone call. Participants will also be reassured that they do not have to take part. The audio-tapes and any printed material relating to the telephone calls will be stored in a secure, locked location before being destroyed in line with the University of Manchester Data Protection Policy. Participants will be asked to propose a convenient date and time for the telephone contact. The researcher will make the call and incur all financial telecommunication charges The telephone contact is expected to last around fifteen minutes, but this estimate may vary depending on how much the participants wish to say.

The interviews and follow-up telephone calls will be audio-taped and transcribed by the researcher, who will ensure any comments that may reveal the identity of a participant are obscured. Anonymising the transcripts in this way preserves participant confidentiality. The researcher will analyse all the data collected during the interviews and telephone calls and code it line by line, allocating the information provided by the participants to relevant themes and categories. This process of analysis will be discussed in the research paper. The researcher will begin to analyse the data soon after conducting the initial interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Participants may be of any gender, ethnicity or socio-economic grouping.
2. Participants must be eighteen years of age or over.
3. Participants must have provided informal, unpaid care or support to a family member, friend or neighbour with dementia during the last twelve months of the life of the person with dementia.

   * This care may have been given on a permanent or intermittent basis.
   * The person with dementia must have died not less than six months and not more than five years prior to the date of the interview.
4. Participants must be able to communicate in English.
5. Participants must have capacity to provide informed consent.
6. Participants must live, or be able to attend an interview, in North West England, West Yorkshire, The West Midlands or North Wales.

Exclusion Criteria:Individuals will be excluded from participating if:

1. They did not give any form of informal unpaid care or support to a person with dementia in the twelve months before that person's death.
2. The person they cared for died less than six months or more than five years before the date of the interview.
3. They are under eighteen years of age.
4. They cannot communicate clearly in English.
5. They are unable or unwilling to provide informed consent.
6. They do not live, or are unable to attend an interview, in North West England, West Yorkshire, the West Midlands or North Wales.
7. The exclusion criteria extend to anyone considered ineligible to approach based on clinical team (Admiral nursing service) concerns about the individual's ability to take part in an interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: family carers of people with dementia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
To conduct interviews with family carers | before 31st December, 2018
  collecting interview data from up to thirty family carers

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No